CLINICAL TRIAL: NCT03626376
Title: A Randomized Trial of Topical Corticosteroid Use in Addition to Oral Antivirals for Prevention of Recurrence of Herpes Simplex Virus (HSV) Keratitis
Brief Title: Topical Corticosteroid Use in Addition to Oral Antivirals for Prevention of Recurrence of Herpes Simplex Virus (HSV) Keratitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to enroll participants
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-01134
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Herpes Simplex Virus Keratitis
MeSH Terms: interventions — Acyclovir; BID protein, human; Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Placebo Comparator): suppressive antiviral treatment
  Interventions: Drug: oral acyclovir 400 mg BID OR valacyclovir 500 mg qdaily
- Study Arm (Active Comparator): oral acyclovir or oral valacyclovir
  Interventions: Drug: oral acyclovir 400 mg BID OR valacyclovir 500 mg qdaily + topical corticosteroid eye drops

INTERVENTIONS:
Drug: oral acyclovir 400 mg BID OR valacyclovir 500 mg qdaily — Treatment used in standard of care
  Arms: Control
Drug: oral acyclovir 400 mg BID OR valacyclovir 500 mg qdaily + topical corticosteroid eye drops — Topical steroid medications to be used in this study include Prednisolone acetate 1.0% or Prednisolone sodium phosphate 1%. The choice of formulation will be dependent on physician preference and medication availability. Formulations of other potencies such as Difluprednate emulsion will not be used in this study. Patients in the study arm will be started on topical corticosteroid 1 drop once a day in the affected eye.
  Arms: Study Arm

SUMMARY:
This is a prospective, randomized clinical trial looking to determine the role of prophylactic treatment with topical corticosteroids in preventing recurrences in patients with a history of infectious epithelial keratitis, stromal keratitis,endotheliitis, or iridocyclitis. Patients will be enrolled to one of two treatment arms: Control arm: oral acyclovir 400 mg BID OR valacyclovir 500 mg daily or Study arm: oral acyclovir 400 mg BID OR valacyclovir 500 mg qdaily + topical corticosteroid eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Subject capable of giving informed consent and if not, an acceptable surrogate capable of giving informed consent on behalf of the subject.
* Diagnosed with a history of herpetic eye disease
* Three or more episodes of HSV keratitis based on medical record documentation of episodes with infectious epithelial keratitis, immune stromal keratitis with or without epithelial ulceration, endothelitis, or iridocyclitis.
* Prior history of HSV keratitis based on medical record documentation of episode of infectious epithelial keratitis, immune stromal keratitis with or without epithelial ulceration, endothelitis, or iridocyclitis and corneal scarring in the central 4mm zone.

Exclusion Criteria:

* Persons who are pregnant or nursing or intend to become pregnant or nurse in the next one year.
* Allergy to acyclovir, fluoromethalone, loteprednol, prednisolone acetate, prednisolone sodium phosphate, or any components of the formulations.
* Persons who are incarcerated.
* Unable to give informed consent or have an acceptable surrogate capable of giving informed consent on behalf of the subject.
* Persons with systemic medical problems who do not agree to have continued medical follow-up.
* History of topical corticosteroids to the eyelids or ocular surface of the involved eye within the prior 30 days prior to enrollment.
* Patients with 3 or more episodes of uveitis in the past 12 months.
* History of keratoplasy or keratorefractive surgery of the involved eye.
* History of open or closed angle glaucoma or ocular hypertension on gtts.
* History of systemic steroid use within the prior 30 days.
* Unable to comply with the study protocol or in the opinion of the investigator would not be a candidate for participation.
* Persons who are unable to instill gtts despite training/caregiver.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-03-02 (Estimated); Study Completion 2022-03-02 (Estimated)

PRIMARY OUTCOMES:
Measure of time to first recurrence | 24 Months
  Kaplan-Meier curves will be plotted by treatment arm (overall and by site) and 95% confidence intervals for the difference between the time to first recurrences will be estimated. Results will also be plotted by site to provide descriptive summaries of the results.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No